CLINICAL TRIAL: NCT06560593
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalation Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics/Pharmacodynamics Characteristics of NTQ5082 Capsules Orally Administered in Healthy Volunteers in Single and Multiple Doses
Brief Title: A Phase 1 Clinical Trial of NTQ5082 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTQ5082-24101
Record Dates: First submitted 2024-07-23; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Complement-mediated Hemolytic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single ascending dose (Experimental): single ascending dose, randomized, double-blind study
  Interventions: Drug: NTQ5082; Drug: Placebo
- multiple ascending dose (Experimental): multiple ascending dose, randomized, double-blind study
  Interventions: Drug: NTQ5082; Drug: Placebo

INTERVENTIONS:
Drug: NTQ5082 — single ascending dose, randomized, double-blind study，with 8 dose groups preset. The first cohort will be the sentinel group, consisted of 2 subjects receiving NTQ5082 capsules. The remaining cohorts required 8 subjects each, with 6 receiving NTQ5082 capsules and 2 receiving placebo.
Drug: Placebo — multiple ascending dose, randomized, double-blind study，with 3 dose groups preset. All cohorts required 8 subjects each, with 6 receiving NTQ5082 capsules and 2 receiving placebo.

SUMMARY:
NTQ5082 capsule is a small molecule CFB factor inhibitor. The study is a randomized, double-blind, placebo-controlled, dose escalation phase 1 clinical trial to evaluate the safety, tolerability and PK/PD characteristics of NTQ5082 capsules orally administered in healthy subjects in single and multiple doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, ≥18 years and ≤45 years in age.
2. 19.0 kg/m2≤BMI≤26.0 kg/m2, and male weight must be ≥50 kg, female weight must be ≥45 kg;
3. Those who sign an informed consent form before the experiment and fully understand the content, process, and possible adverse reactions of the experiment;
4. The subjects are able to communicate well with the researchers and understand and comply with the requirements of this study.

3. (Part 2 only) The Subjects voluntarily receive ACYW135 group meningococcal vaccine and pneumococcal vaccine at least 14 days before NTQ5082 capsule administration. If the subjects has received pneumococcal vaccine within 5 years, or ACYW135 group meningococcal vaccine within 3 years, repeated vaccination is not required.

Exclusion Criteria:

1. Participants who have participated in any other drug clinical trials and used the investigational drug within 3 months prior to the trial;
2. Individuals who have chronic or active gastrointestinal diseases such as esophageal disease, gastritis, gastric ulcer, gastroesophageal reflux, enteritis, active gastrointestinal bleeding, or gastrointestinal surgery within the past three years, and who are still clinically significant according to researchers;
3. Individuals with clear diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, metabolic disorders, etc. that require medical intervention or other diseases that are not suitable for clinical trials (such as a history of mental illness);
4. Known or suspected history of immunodeficiency (such as frequent recurrent infections), genetic or acquired complement deficiency;
5. There is a clear history of capsule microbial infection within the first 6 months of screening; Including but not limited to: history of infection with Streptococcus pneumoniae, Bacillus anthracis, Salmonella, Salmonella typhi, Klebsiella pneumoniae, Pseudomonas aeruginosa, Bacteroides fragilis, Neisseria meningitidis, Haemophilus influenzae, Legionella pneumophila;
6. Individuals with a history of tuberculosis infection or currently suffering from tuberculosis infection;
7. Active systemic bacterial, viral, or fungal infection within 14 days prior to administration;
8. Fever (≥ 38 ℃) occurred within 7 days before administration;
9. Individuals with a history of allergies to experimental preparations, any of their components or related preparations, or to drugs, food or other substances;
10. Those who cannot tolerate venous puncture or have a history of dizziness or needle fainting;
11. Patients who have undergone surgery within 6 months prior to the use of the investigational drug, as determined by the researcher, that may affect drug absorption, distribution, metabolism, and excretion; Or have undergone surgical procedures within 4 weeks prior to using the investigational drug; Or those who plan to undergo surgical procedures during the trial period;
12. Those who have used any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, traditional Chinese patent medicines and simple preparations and dietary supplements) within 2 weeks before using the study drug; Or screen for drugs with a duration of less than 5 half lives (whichever is longer);
13. Individuals who have received the vaccine or live attenuated vaccine within 14 days prior to using the investigational drug, or who plan to receive the vaccine during the trial period;
14. Individuals with QTc>450 milliseconds (male) or QTc>470 milliseconds (female) during screening;
15. Individuals who have donated blood or experienced significant blood loss (>400mL) within 3 months prior to the use of the investigational drug, those who have received blood transfusions or used blood products, or those who intend to donate blood or blood components during or within 3 months after the end of the trial;
16. Drug abusers or those who have used soft drugs (such as marijuana) or hard drugs (such as cocaine, phencyclidine, etc.) within the past year before using research drugs; Or those who test positive for urinary toxicity screening;
17. Smokers or those who have smoked more than 5 cigarettes per day in the 3 months prior to using the study drug, or those who cannot stop using any tobacco products during the trial period;
18. Alcoholics or frequent drinkers within the 6 months prior to the experiment, who consume more than 14 units of alcohol per week (1 unit=360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); Those who are unwilling to stop drinking alcohol or any alcoholic products during the trial period; Or those who test positive for alcohol breath test;
19. Individuals who consume excessive amounts of tea, coffee, and/or caffeinated beverages (8 or more cups, 1 cup=250 mL) daily, or who do not agree to stop drinking tea, coffee, and/or caffeinated beverages during the trial period;
20. Individuals who consume a diet (including grapefruit or grapefruit products, etc.) that may affect the metabolism of the investigational drug within 7 days prior to use, or who are deemed by the researcher to have other diets that may affect the absorption, distribution, metabolism, or excretion of the drug, or who do not agree to stop consuming the aforementioned foods during the trial period;
21. Those who have special dietary requirements and cannot follow a uniform diet;
22. Female subjects are pregnant or breastfeeding women; Or engaging in unprotected sexual activity within 2 weeks prior to the use of the investigational drug; Those who have used oral contraceptives within 30 days prior to the use of the study drug, or those who have used long-acting estrogen or progesterone injections or implants within 6 months prior to the use of the study drug;
23. If the subject (or their partner) has a pregnancy plan, sperm and egg donation plan, or is unwilling to take one or more non pharmacological contraceptive measures (such as complete abstinence, contraceptive rings, partner ligation, etc.) within 3 months after the last dose of medication from the time of signing the informed consent form;
24. Physical examination, electrocardiogram, abdominal ultrasound, chest radiograph, laboratory tests (blood routine, reticulocyte count, procalcitonin, high-sensitivity C-reactive protein, urine routine, blood biochemistry, thyroid function, coagulation function, D-dimer, blood transfusion, blood pregnancy), vital signs, and clinically significant abnormalities in various examinations (subject to the judgment of the research doctor);
25. Participants may not be able to complete this study due to other reasons or may have other reasons deemed inappropriate by the researchers to participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
the safety and tolerability | up to 21 days
  Safety and tolerability as assessed through collection of Adverse Event, Serious Adverse Event, Clinical Chemistry/Haematology/Coagulation/Vital Signs and ECG

SECONDARY OUTCOMES:
AUC0-last in plasma of part 1 | up to 11 days
AUC0-∞ in plasma of part 1 | up to 11 days
Cmax in plasma of part 1 | up to 11 days
Tmax in plasma of part 1 | up to 11 days
t1/2 in plasma of part 1 | up to 11 days
Aet1-t2 in urine of part 1 | up to 11 days
Ae0-t in urine of part 1 | up to 11 days
Fe0-t in urine of part 1 | up to 11 days
CLr in urine of part 1 | up to 11 days
AUC0-τ in plasma after the first dosing of part 2 | up to 21 days
AUC0-∞ in plasma after the first dosing of part 2 | up to 21 days
Tmax in plasma after the first dosing of part 2 | up to 21 days
Cmax in plasma after the first dosing of part 2 | up to 21 days
AUC0-τ,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days
AUC0-t,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days
AUC0-∞,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days
Tmax,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days
Cmax,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days
Ctrough,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days
Cavg,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days
t1/2,ss in plasma under steady-state conditions (ss) of part 2 | up to 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Third hospital of Changsha, Changsha, Hunan, China